CLINICAL TRIAL: NCT02055703
Title: A 3-Part, Open-Label, Drug-Drug Interaction Study of Concomitant Administration of E2609 With Itraconazole, Rifampin, Digoxin, or Donepezil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2609-A001-003
Record Dates: First submitted 2014-01-23; First posted 2014-02-05 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects
MeSH Terms: interventions — Itraconazole; Rifampin; Digoxin; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- E2609 (Experimental): Experimental drug for Parts A, B, and C
  Interventions: Drug: itraconazole; Drug: rifampin; Drug: digoxin; Drug: donepezil
- itraconazole (Active Comparator): Comparator drug for Part A1
  Interventions: Drug: E2609
- rifampin (Active Comparator): Comparator drug for Part A2
  Interventions: Drug: E2609
- digoxin (Active Comparator): Comparator drug for Part B
  Interventions: Drug: E2609
- donepezil (Active Comparator): Comparator drug for Part C
  Interventions: Drug: E2609

INTERVENTIONS:
Drug: E2609
  Arms: digoxin; donepezil; itraconazole; rifampin
Drug: itraconazole
  Arms: E2609
Drug: rifampin
  Arms: E2609
Drug: digoxin
  Arms: E2609
Drug: donepezil
  Arms: E2609

SUMMARY:
This study will be a single-center, open-label, drug-drug interaction study in healthy male and female subjects. The study will consist of 3 parts: A, B, and C. In Part A, the effect of itraconazole or rifampin on the pharmacokinetics (PK) of E2609 and metabolites will be assessed. Approximately 32 subjects will be assigned to 1 of 2 treatment groups (itraconazole or rifampin) in equal numbers, with approximately 16 subjects per group. In Part B, the effects of steady-state dosing of E2609 on the PK of digoxin will be assessed in approximately 18 subjects. In Part C, the effects of donepezil administered in combination with, or 2 hours after, E2609 dosing on the PK of E2609 and metabolites, will be assessed in approximately 24 subjects.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male or female subjects aged 18-55 years inclusive at the time of informed consent
2. Provide written informed consent
3. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

1. Any history of seizures or epilepsy (not including a history of simple febrile seizures in childhood) or disturbance of consciousness likely to be due to seizures
2. A prolonged QT/QTc interval (QTc greater than 450 ms) as demonstrated by the mean of triplicate electrocardiograms (ECGs), recorded at least 1 min apart, at Screening or Baseline Periods
3. Evidence of clinically significant disease (eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system) that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments or subjects who have a congenital abnormality in metabolism within 4 weeks before dosing.
4. Any laboratory abnormalities considered clinically significant by the investigator, which may require further investigations or treatment
5. Clinically significant illness which required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of single oral doses of E2609 and metabolites in subjects dosed alone or in combination with either rifampin or itraconazole | Up to 48 days (Part A)
  Primary PK Parameters being measured: AUC(0-t), AUC(0-inf), Cmax, tmax.
To evaluate the PK of single oral doses of digoxin in subjects dosed alone or in combination with E2609 | Up to 48 days (Part B)
  Primary PK Parameters being measured: AUC(0-t), AUC(0-inf), Cmax, tmax.
To evaluate the PK of single oral doses of E2609 and metabolites in subjects dosed alone, in combination with donepezil, or 2 hours before donepezil dosing | Up to 86 day (Part C)
  Primary PK Parameters being measured: AUC(0-t), AUC(0-inf), Cmax, tmax.

SECONDARY OUTCOMES:
Safety and tolerability of single oral doses of E2609 in subjects in the presence and absence of rifampin, itraconazole, digoxin, or donepezil | Up to 182 days
  Safety assessments include monitoring and recording all adverse events (AEs), regular measurement of vital signs, and the performance of physical examinations.
To evaluate the effects of DNA sequence variants potentially involved in absorption, distribution and metabolism of E2609. | Up to 182 days
  DNA samples will be collected, stored, and may be used to examine the role of genetic variability in other genes potentially involved in absorption, distribution, metabolism, and excretion.

CONTACTS AND LOCATIONS:
Locations (1):
- WCT Early Development, San Antonio, Texas, United States